CLINICAL TRIAL: NCT06408727
Title: An Intermediate Expanded Access Protocol With CNM-Au8 for Amyotrophic Lateral Sclerosis for NIH Grant RFA-NS-23-012
Brief Title: Intermediate Expanded Access Protocol CNMAu8.EAP04
Status: Available | Type: Expanded Access
Sponsor: Clene Nanomedicine (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: CNMAu8.EAP04; 1U01NS136023-01 (NIH)
Record Dates: First submitted 2024-04-24; First posted 2024-05-10 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: ALS; Amyotrophic Lateral Sclerosis; PALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: CNM-Au8 — CNM-Au8 (cellular energetic nanocatalyst). Faceted clean-surfaced catalytically-active Au nanocrystals.

SUMMARY:
An Intermediate Expanded Access Protocol (EAP) with CNM-Au8 for Amyotrophic Lateral Sclerosis for NIH Grant RFA-NS-23-012

DETAILED DESCRIPTION:
An Intermediate Expanded Access Protocol (EAP) with CNM-Au8 for Amyotrophic Lateral Sclerosis for NIH Grant RFA-NS-23-012. The primary objective of this intermediate EAP is to provide access to the investigational product, CNM-Au8 30mg, for up to 180 people living with ALS.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give written informed consent.
2. Male or female participants aged 18 years or greater (inclusive) at the time of informed consent completion.
3. Participants with a confirmed diagnosis of ALS per Gold Coast criteria as determined by a neurologist specializing in ALS (e.g., the site principal investigator or sub-investigator for this study).
4. Participant is able to daily consume up to 60 mL of the investigational drug suspension without substantial dysphagia, OR can intake the investigational product through a feeding tube.
5. Participant must have completed standard clinical safety labs within the prior 90 days from the Baseline visit, including a chemistry panel (e.g., CMP) and a hematology panel (e.g., CBC).
6. Participant has a baseline score by the TRICALS risk calculator that is less than -2 (i.e., participant is not at increased risk of early death; https://tricals.shinyapps.io/risk-profile/).
7. Participant meets the following criteria:

   1. Baseline Vital Capacity >15% predicted,
   2. Baseline ALSFRS-R Score >8, and,
   3. Baseline BMI >17.5 kg/m2
8. Participants have established care with a neurologist at the specialized ALS center or remotely enrolling site involved in the study and will maintain this clinical care throughout the duration of the EAP within the United States.

Exclusion Criteria:

1. Participant is eligible for participation in any double-blind placebo-controlled study the treatment of ALS at the same research site.
2. Participant has a history of any clinically significant or unstable medical condition (other than ALS) that may interfere with assessment of safety or compromise the study objectives.
3. Based on the investigator's judgment, participants who may have difficulty complying with the protocol and/or any study procedures.
4. Within the prior 90-days the participant has had clinically significant findings on standard hepatic, hematologic, or renal safety assays, including but not limited to: (i) ALT or AST ≥ 3 times upper limits of normal, (ii) direct (conjugated) with bilirubin ≥2 times upper limits of normal, (iii) low platelet counts (< 150 x 109 per liter) or eosinophilia (absolute eosinophil count of ≥ 500 eosinophils per microliter), (iv) serum creatinine >1.2 mg/dL, or (v) eGFR < 45 ml/min per 1.73 m2.
5. Participant is currently involved in another placebo-controlled clinical trial (note: concomitant therapy with other investigational products is permitted with certain restrictions-see concomitant medications below).
6. Females who are pregnant or nursing or who plan to get pregnant during the EAP, or within 6 months of the end of this trial.
7. Females of child-bearing potential, or men, who are unwilling or unable to use accepted methods of birth control.
8. History of gold allergy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Northwestern University, Chicago, Illinois
  - Synapticure, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Columbia Unniversity, New York, New York
  - Duke University, Durham, North Carolina
  - Pennsylvania State University, Hershey, Pennsylvania
  - Texas Neurology, Dallas, Texas